CLINICAL TRIAL: NCT05343390
Title: Enhancing HIV-assisted Contact Tracing in Malawi Through Blended Learning: an Implementation Science Study
Brief Title: Package of Resources for Assisted Contact Tracing: Implementation, Costs, and Effectiveness
Acronym: PRACTICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-1810; R01MH124526 (NIH)
Record Dates: First submitted 2022-04-08; First posted 2022-04-25 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: blended learning; digital learning; quality improvement; HIV testing; health care worker capacity building
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized control trial with 2:1 randomization (standard: enhanced).
Who Masked: Outcomes Assessor
Masking Description: Participants and investigators will not be masked. For fidelity assessments, those coding audio recordings will be masked with respect to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced implementation strategy (Experimental): digitally guided training and continuous quality improvement
  Interventions: Behavioral: Enhanced implementation package; Behavioral: Standard implementation package
- Standard implementation strategy (Active Comparator): standard training and clinical support
  Interventions: Behavioral: Standard implementation package

INTERVENTIONS:
Behavioral: Enhanced implementation package — Individual training with teaching and modeling (tablet-guided, ~8 hours) Small group training with practice and feedback (tablet-guided, ~16 hours) Ongoing continuous quality improvement sessions (tablet-guided, ~2 hours/month)
  Arms: Enhanced implementation strategy
Behavioral: Standard implementation package — Individual training with teaching (facilitator-guided, ~2 hours) Small group practice (facilitator-guided, ~1 hour) Ongoing clinic support (facilitator-guided, ~30 minutes/month)

SUMMARY:
Having health workers assist HIV-infected persons with the recruitment and testing of their sexual contacts and biological children is an effective and efficient way of identifying additional HIV-infected persons in need of HIV treatment and HIV-uninfected persons in need of HIV prevention. However, in Malawi, a country with a generalized HIV epidemic, health workers lack the counseling and coordination skills to routinely assist their HIV-infected clients with these services. This study will determine how to help health workers to effectively and efficiently provide these services to their patients through a set of digital capacity-building tools.

DETAILED DESCRIPTION:
Voluntary assisted contact tracing (ACT) is an evidence-based approach that efficiently identifies persons in need of HIV treatment and prevention. Malawi, like many countries in sub-Saharan Africa, has adopted ACT policies to support its "95-95-95" targets for HIV testing, treatment, and viral suppression.

However, Malawi's ACT implementation has been poor due to deficits in health worker capacity and clinical coordination. Through preliminary work, our team has 1) developed a set of implementation strategies (theory-based health worker training and continuous quality improvement processes) that address these barriers; 2) packaged these strategies into a blended learning platform that combines digital and face-to-face modalities; and 3) field-tested the package in Malawi with promising preliminary results. In this proposal, the package will be rigorously evaluated in Malawi for implementation, service uptake, and cost-effectiveness outcomes.

Through a two-arm pragmatic cluster randomized implementation trial, the proposed research will address these gaps through three specific aims. Twenty Malawian facilities in two districts will be randomized to receive the blended learning implementation package (enhanced) versus standard implementation package (standard). In the first aim, ACT implementation outcomes will be compared between the enhanced and standard arms. Health worker fidelity to ACT procedures will be assessed through audio-recorded ACT encounters. In the second aim, HIV service uptake outcomes will be compared between the enhanced and standard arms. In the third aim, cost and cost-effectiveness outcomes will be examined.

The findings will offer important insights and innovations into how to bridge the gap between ACT research and practice, a critical step towards achieving the 95-95-95 targets.

ELIGIBILITY:
Health worker inclusion criteria:

* 18 years of age or older
* working full-time at one of the health facilities included in the study
* staff in Malawi's Assisted Contact Tracing program.

Health worker exclusion criteria:

* conditions that would compromise ability of participant to provide informed consent, undergo study procedures safely, or prevent proper conduct of study

Patient (index or contact) inclusion criteria:

->=15 years

-potential index, contact, or parent or guardian of a potential index or contact

Patient (index or contact) exclusion criteria:

* conditions that would compromise ability of individual to provide informed consent, undergo study procedures safely, or prevent proper conduct of study

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Rosenberg, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (33):
- Malawi (33):
  - Balaka District Hospital, Balaka
  - Balaka OPD Health Centre, Balaka
  - Chiendausiku Health Centre, Balaka
  - Kalembo Health Centre, Balaka
  - Kankao Health Centre, Balaka
  - Kwitanda Health Centre, Balaka
  - Mbera Health Centre, Balaka
  - Namanolo Health Centre, Balaka
  - Namdumbo Health Centre, Balaka
  - Phalula Health Centre, Balaka
  - Phimbi Health Centre, Balaka
  - Ulongwe Health Centre, Balaka
  - Utale Health Centres, Balaka
  - Chamba Dispensary, Machinga
  - Chikweo Health Centre, Machinga
  - Gawanani Health Centre, Machinga
  - Kawinga Dispensary, Machinga
  - Machinga District Hospital, Machinga
  - Mahinga Health Centre, Machinga
  - Mangamba Health Centre, Machinga
  - Mbonechela Dispensary, Machinga
  - Mkwepere Health Centre, Machinga
  - Mpiri Health Centre, Machinga
  - Mposa Health Centre, Machinga
  - Namandanje Health Centre, Machinga
  - Namanja Health Centre, Machinga
  - Nayinunje Health Centre, Machinga
  - Nayuchi Health Centre, Machinga
  - Ngokwe health Centre, Machinga
  - Nsanama Health Centre, Machinga
  - Ntaja Health Centre, Machinga
  - Nthorowa Health Centre, Machinga
  - Nyambi Health Centre, Machinga

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, all data will be de-identified and shared in compliance with all regulatory bodies and NIH data sharing procedures.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months after publication and continuing through 36 months of publication
Access Criteria: A repository will be selected that has policies and procedures in place that will provide data access to qualified researchers, fully consistent with NIH data sharing policies and applicable laws and regulations. The researcher will need approval form an Institutional Review Board and an executed data use/sharing agreement with University of North Carolina at Chapel Hill investigators.

REFERENCES:
- [Derived] Meek CJ, Munkhondya TEM, Mphande M, Tembo TA, Chitani M, Jean-Baptiste M, Vansia D, Kumbuyo C, Wang J, Simon KR, Rutstein SE, Barrington C, Kim MH, Go VF, Rosenberg NE. Examining the feasibility of assisted index case testing for HIV case-finding: a qualitative analysis of barriers and facilitators to implementation in Malawi. BMC Health Serv Res. 2024 May 9;24(1):606. doi: 10.1186/s12913-024-10988-z. PMID 38720312
- [Derived] Tembo TA, Mollan K, Simon K, Rutstein S, Chitani MJ, Saha PT, Mbeya-Munkhondya T, Jean-Baptiste M, Meek C, Mwapasa V, Go V, Bekker LG, Kim MH, Rosenberg NE. Does a blended learning implementation package enhance HIV index case testing in Malawi? A protocol for a cluster randomised controlled trial. BMJ Open. 2024 Jan 22;14(1):e077706. doi: 10.1136/bmjopen-2023-077706. PMID 38253452
- [Derived] Meek CJ, Munkhondya TEM, Mphande M, Tembo TA, Chitani M, Jean-Baptiste M, Vansia D, Kumbuyo C, Simon KR, Rutstein SE, Barrington C, Kim MH, Go VF, Rosenberg NE. Examining the feasibility of assisted index case testing for HIV case-finding: a qualitative analysis of barriers and facilitators to implementation in Malawi. Res Sq [Preprint]. 2023 Sep 8:rs.3.rs-3314925. doi: 10.21203/rs.3.rs-3314925/v1. PMID 37720011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 clusters were randomized in a 1:2 ratio (Enhanced:Standard). Within these clusters Healthcare workers, Index clients, Contact clients and data from registers were observed. To clearly represent the groups within each arm, four "periods" are shown below. Periods do not reflect a time element, but rather the four populations measured within these clusters (units).
Units Other Than Participants: Clusters
Period: Clusters and Healthcare Workers
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Started | 125; 11 Clusters | 181; 22 Clusters
Completed | 115; 11 Clusters | 174; 22 Clusters
Not Completed | 10; 0 Clusters | 7; 0 Clusters
Period: Clusters and Index Clients
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Started | 124; 11 Clusters | 217; 22 Clusters
Completed | 124; 11 Clusters | 217; 22 Clusters
Not Completed | 0; 0 Clusters | 0; 0 Clusters
Period: Clusters and Contact Clients
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Started | 67; 11 Clusters | 127; 22 Clusters
Completed | 67; 11 Clusters | 127; 22 Clusters
Not Completed | 0; 0 Clusters | 0; 0 Clusters
Period: Clusters and Register-Extracted Data
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Started | 21248; 11 Clusters | 33272; 22 Clusters
Completed (The Cluster and Register-Extracted data are not considered enrolled participants in the study. These de-identified data were extracted from registers in aggregate and no data were collected directly from these individuals.) | 21248; 11 Clusters | 33272; 22 Clusters
Not Completed | 0; 0 Clusters | 0; 0 Clusters

BASELINE CHARACTERISTICS:
Population: In the Enhanced arm there were 125 Healthcare workers, 124 index clients, and 67 contact clients for a total of 316. In the Standard arm, there were 181 Healthcare workers, 217 Index clients, and 127 Contact clients for a total of 525. The "Cluster and Register-Extracted data" population were not considered as enrolled participants in the study; they were extracted data from register and no data were collected from these individuals.
Groups:
- Enhanced Implementation Strategy: Standard training and clinical support
  + Enhanced digitally guided training and continuous quality improvement
- Total: Total of all reporting groups
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy | Total
Number analyzed (Participants) | 316 | 525 | 841
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Data are reported separately for Heathcare Workers, Index clients, and Contact clients. Data were not provided by 1 healthcare worker.
  years
    Healthcare Workers: number analyzed (Participants) | 125 | 180 | 305
    Healthcare Workers | 34 [28 to 38] | 33 [27 to 40] | 34 [28 to 39]
    Index Clients: number analyzed (Participants) | 124 | 217 | 341
    Index Clients | 35 [27 to 40] | 34 [27 to 40] | 34 [27 to 42]
    Contact Clients: number analyzed (Participants) | 67 | 127 | 194
    Contact Clients | 39 [30 to 48] | 35 [29 to 45] | 37 [29 to 47]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data are reported separately for Heathcare Workers, Index clients, and Contact clients.
  Participants
    Healthcare Workers: number analyzed (Participants) | 125 | 180 | 305
    Healthcare Workers: Female | 59 | 87 | 146
    Healthcare Workers: Male | 66 | 93 | 159
    Index Clients: number analyzed (Participants) | 124 | 217 | 341
    Index Clients: Female | 81 | 159 | 240
    Index Clients: Male | 43 | 58 | 101
    Contact Clients: number analyzed (Participants) | 67 | 127 | 194
    Contact Clients: Female | 25 | 61 | 86
    Contact Clients: Male | 42 | 66 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Heathcare Workers, Index clients, and Contact clients.
  Participants
    Healthcare Workers: number analyzed (Participants) | 125 | 181 | 306
    Healthcare Workers: Hispanic or Latino | 0 | 0 | 0
    Healthcare Workers: Not Hispanic or Latino | 123 | 181 | 304
    Healthcare Workers: Unknown or Not Reported | 2 | 0 | 2
    Index Clients: number analyzed (Participants) | 124 | 217 | 341
    Index Clients: Hispanic or Latino | 0 | 0 | 0
    Index Clients: Not Hispanic or Latino | 124 | 217 | 341
    Index Clients: Unknown or Not Reported | 0 | 0 | 0
    Contact Clients: number analyzed (Participants) | 67 | 127 | 194
    Contact Clients: Hispanic or Latino | 0 | 0 | 0
    Contact Clients: Not Hispanic or Latino | 67 | 127 | 194
    Contact Clients: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data are reported separately for Heathcare Workers, Index clients, and Contact clients.
  Participants
    Healthcare Workers: number analyzed (Participants) | 125 | 180 | 305
    Healthcare Workers: American Indian or Alaska Native | 0 | 0 | 0
    Healthcare Workers: Asian | 0 | 0 | 0
    Healthcare Workers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Healthcare Workers: Black or African American | 125 | 180 | 305
    Healthcare Workers: White | 0 | 0 | 0
    Healthcare Workers: More than one race | 0 | 0 | 0
    Healthcare Workers: Unknown or Not Reported | 0 | 0 | 0
    Index Clients: number analyzed (Participants) | 124 | 217 | 341
    Index Clients: American Indian or Alaska Native | 0 | 0 | 0
    Index Clients: Asian | 0 | 0 | 0
    Index Clients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Index Clients: Black or African American | 124 | 217 | 341
    Index Clients: White | 0 | 0 | 0
    Index Clients: More than one race | 0 | 0 | 0
    Index Clients: Unknown or Not Reported | 0 | 0 | 0
    Contact Clients: number analyzed (Participants) | 67 | 127 | 194
    Contact Clients: American Indian or Alaska Native | 0 | 0 | 0
    Contact Clients: Asian | 0 | 0 | 0
    Contact Clients: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Contact Clients: Black or African American | 67 | 127 | 194
    Contact Clients: White | 0 | 0 | 0
    Contact Clients: More than one race | 0 | 0 | 0
    Contact Clients: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 316 | 525 | 841

OUTCOME MEASURES:

1. Primary Outcome: Index Client Fidelity Assessment
Description: Health care workers will be observed counseling actual index clients. The scores on the 15-item index client fidelity assessment will be compared between arms (range 0-100% with higher scores being better)
Time Frame: 1 year after training
Population: Data were missing for 2 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 122 | 217
score on a scale | 66.30 [62.8 to 69.7] | 45.70 [42.8 to 48.6]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p < 0.001, Regression, Linear; A linear model fit using generalized estimating equations to account for correlated observations within clusters; Mean Difference (Final Values) = 20.6, 95% CI 2-sided [16.1 to 25.1]

2. Primary Outcome: Contact Client Fidelity Assessment
Description: Health care workers will be observed counseling actual contact clients. The scores on the 15-item contact client fidelity assessment will be compared between arms (range 0-100% with higher scores being better)
Time Frame: 1 year after training
Population: Data were missing for 3 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 64 | 127
score on a scale | 63.70 [58.8 to 68.6] | 52.50 [50.8 to 54.2]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p < 0.001, Regression, Linear; A linear model fit using generalized estimating equations to account for correlated observations within clusters; Mean Difference (Final Values) = 11.1, 95% CI 2-sided [5.9 to 16.4]

3. Primary Outcome: Index Clients Who Participate in Assisted Contact Tracing
Description: The total number of index clients who participate in assisted contact tracing relative to the number of total potential index clients measured per facility per calendar quarter (3-month period). Each cluster contributes 4 quarters of data.
Time Frame: 1 year after training
Population: Data unavailable for one cluster in Quarter 4 of the standard arm.
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Units Other Than Participants: Cluster-quarters
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 21248 | 33272
Number analyzed (Cluster-quarters) | 44 | 87
proportion of participants | 0.56 [0.33 to 0.87] | 0.46 [0.30 to 0.68]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p = 0.14, Mixed Models Analysis; Negative binomial mixed-effect model; Rate Ratio = 1.22, 95% CI 2-sided [0.93 to 1.60]

4. Primary Outcome: Contact Clients Elicited
Description: The number of contact clients listed by participating index clients relative to the number of total potential index clients measured per facility per calendar quarter (3-month period). Each cluster contributes 4 quarters of data.
Time Frame: 1 year after training
Population: Data unavailable for one cluster in Quarter 4 of the standard arm.
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Units Other Than Participants: Cluster-quarters
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 21248 | 33272
Number analyzed (Cluster-quarters) | 44 | 87
proportion of participants | 0.19 [0.13 to 0.27] | 0.13 [0.09 to 0.19]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p = 0.006, Mixed Models Analysis; Negative binomial mixed-effect model; Rate Ratio = 1.37, 95% CI 2-sided [1.10 to 1.71]

5. Primary Outcome: HIV Self-test Kits Distributed
Description: The number of HIV self-test kits distributed relative to the number of total potential index clients measured per facility per calendar quarter (3-month period). Each cluster contributes 4 quarters of data.
Time Frame: 1 year after training
Population: Data unavailable for one cluster in Quarter 4 of the standard arm.
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Units Other Than Participants: Cluster-quarters
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 21248 | 33272
Number analyzed (Cluster-quarters) | 44 | 87
proportion of participants | 0.016 [0.008 to 0.028] | 0.006 [0.000 to 0.016]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p = 0.013, Mixed Models Analysis; Negative binomial mixed-effect model; Rate Ratio = 2.29, 95% CI 2-sided [1.19 to 4.40]

6. Primary Outcome: Contact Clients Tested
Description: The number of contact clients tested relative to the number of total potential index clients measured per facility per calendar quarter (3-month period). Each cluster contributes 4 quarters of data.
Time Frame: 1 year after training
Population: Data unavailable for one cluster in Quarter 4 of the standard arm.
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Units Other Than Participants: Cluster-quarters
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 21248 | 33272
Number analyzed (Cluster-quarters) | 44 | 87
proportion of participants | 0.11 [0.06 to 0.20] | 0.08 [0.05 to 0.11]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p = 0.01, Mixed Models Analysis; Negative binomial mixed-effect model; Rate Ratio = 1.45, 95% CI 2-sided [1.10 to 1.92]

7. Primary Outcome: Contact Clients Living With HIV Identified
Description: The number of contact clients living with HIV identified relative to the number of total potential index clients measured per facility per calendar quarter (3-month period). Each cluster contributes 4 quarters of data.
Time Frame: 1 year after training
Population: Data unavailable for one cluster in Quarter 4 of the standard arm.
Measure: Median (Inter-Quartile Range); unit: proportion of participants
Units Other Than Participants: Cluster-quarters
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 21248 | 33272
Number analyzed (Cluster-quarters) | 44 | 87
proportion of participants | 0.005 [0.002 to 0.008] | 0.004 [0.003 to 0.008]
Statistical Analysis 1: Comparison: Enhanced Implementation Strategy vs Standard Implementation Strategy; Test type: Superiority; p = 0.12, Mixed Models Analysis; Negative binomial mixed-effect model; Rate Ratio = 1.28, 95% CI 2-sided [0.94 to 1.76]

8. Primary Outcome: Incremental Cost Per Contact Tested
Description: Incremental cost per contact tested for HIV = Total additional cost in enhanced arm ($127,319) / total number of additional individual tested for HIV in the enhanced arm (1119). The outcome is an incremental cost effectiveness ratio. Because no additional cost was incurred in the Standard arm, the value was reported as 0.
Time Frame: 1 year after training
Population: Calculations were driven from the 'Clusters and Register-Extracted Data' population. The full range of incremental cost was derived based on variability in cost associated with implementation strategy development. Number of participants analyzed in the Standard Arm is Zero due to this outcome being an incremental measure; no additional clients were tested in the Standard Arm.
Measure: Mean (Full Range); unit: US Dollars
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 1119 | 0
US Dollars | 114 [70 to 142] |

9. Primary Outcome: Incremental Cost Per Person Living With HIV Diagnosed
Description: Incremental cost per contact tested for HIV = Total additional cost in enhanced arm ($127,319) / total number of additional individual diagnosed with HIV in the enhanced arm (64). The outcome is an incremental cost effectiveness ratio. Because no additional cost was incurred in the Standard arm, the value is reported as 0.
Time Frame: 1 year after training
Population: Calculations were driven from the 'Clusters and Register-Extracted Data' population. The full range of incremental cost was derived based on variability in cost associated with implementation strategy development. Number of participants analyzed in the Standard Arm is Zero due to this outcome being an incremental measure; no additional clients were diagnosed with HIV in the Standard Arm.
Measure: Mean (Full Range); unit: US Dollars
Arm/Group | Enhanced Implementation Strategy | Standard Implementation Strategy
Number analyzed (Participants) | 64 | 0
US Dollars | 1977 [1209 to 2471] |

ADVERSE EVENTS:
Time Frame: From the time of enrollment through study completion (approximately 12 months).
Description: The "Cluster and Register-Extracted data" population are not considered enrolled participants in the study. These are extracted data from register and no data were collected from these individuals.
Groups:
- Enhanced Implementation Strategy Healthcare Workers; Enhanced Implementation Strategy Index Clients; Enhanced Implementation Strategy Contact Clients: Standard training and clinical support
  + Enhanced digitally guided training and continuous quality improvement
- Standard Implementation Strategy Healthcare Workers; Standard Implementation Strategy Index Clients; Standard Implementation Strategy Contact Clients: Standard training and clinical support
Arm/Group | Enhanced Implementation Strategy Healthcare Workers | Enhanced Implementation Strategy Index Clients | Enhanced Implementation Strategy Contact Clients | Standard Implementation Strategy Healthcare Workers | Standard Implementation Strategy Index Clients | Standard Implementation Strategy Contact Clients
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/124 | 0/67 | 1/181 | 0/217 | 0/127
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/124 | 0/67 | 1/181 | 0/217 | 0/127
Other Adverse Events (participants affected / at risk) | 0/125 | 0/124 | 0/67 | 0/181 | 0/217 | 0/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Implementation Strategy Healthcare Workers (N=125) | Enhanced Implementation Strategy Index Clients (N=124) | Enhanced Implementation Strategy Contact Clients (N=67) | Standard Implementation Strategy Healthcare Workers (N=181) | Standard Implementation Strategy Index Clients (N=217) | Standard Implementation Strategy Contact Clients (N=127)
Surgery complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05343390/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05343390/ICF_000.pdf